CLINICAL TRIAL: NCT02283216
Title: Acoustic Stimulation Paired With Body and Cortical Stimulation for Modulating Tinnitus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding and personnel
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1409M53708
Record Dates: First submitted 2014-10-26; First posted 2014-11-05 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Tinnitus
Keywords: neuromodulation; noninvasive; plasticity; transcranial magnetic stimulation; hearing; hyperacusis
MeSH Terms: conditions — Tinnitus; Hyperacusis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acoustic, Body, Cortical (Experimental): Acoustic corresponds to noise sound stimulation. Body corresponds to body electrical stimulation. Cortical corresponds to transcranial magnetic stimulation. Acoustic is presented together with body and cortical stimulation. Different body locations and timing among acoustic, body, and cortical stimulation are presented across testing sessions.
  Interventions: Device: noise sound stimulation (Tucker-Davis Technologies); Device: body electrical stimulation (Digitimer device); Device: transcranial magnetic stimulation (Magstim)

INTERVENTIONS:
Device: noise sound stimulation (Tucker-Davis Technologies) — Band-limited white noise stimulus, comfortable loudness level, presented via headphones or earphones with Tucker-Davis Technologies device.
Device: body electrical stimulation (Digitimer device) — Single pulse electrical stimulation on different body regions, comfortable current level, presented via surface pads or clips with Digitimer device.
Device: transcranial magnetic stimulation (Magstim) — Single pulse magnetic stimulation over frontal cortex, comfortable level at 110% resting motor threshold, presented via magnetic coil with Magstim device.

SUMMARY:
The purpose of the study is to investigate different stimulation parameters for a new noninvasive approach for modulating the brain that could potentially be beneficial for decreasing tinnitus perception. The new approach is called Multimodal Synchronization Therapy (mSync). mSync uses a combination of acoustic stimulation played through headphones and low levels of electrical current delivered via electrodes placed on the surface of different body regions. The timing interval between the acoustic and body stimulation is varied in order to cause different types of changes in the brain. In addition to acoustic and body stimulation, noninvasive cortical stimulation will also be presented as part of mSync to attempt to further modulate or decrease the tinnitus percept. Cortical stimulation will be performed by placing a magnetic coil over a spot on the head and sending a brief magnetic pulse that can travel through the skin and bone to create electrical current inside the head. For this study, different body locations as well as specific timing intervals among acoustic, body, and cortical stimulation will be investigated to identify appropriate parameters that can modulate and potentially decrease tinnitus perception. Different mSync parameters will be investigated across multiple testing sessions (up to 16 weekly sessions) and the tinnitus percept will be closely monitored throughout the study.

DETAILED DESCRIPTION:
This study is not specifically seeking to treat tinnitus but is designed to investigate various mSync parameters that can alter the tinnitus percept. Findings from this study will help identify specific mSync parameters that can be more effective at decreasing or fully suppressing the tinnitus percept that will be systematically explored in a follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Have subjective, non-pulsatile, and bothersome tinnitus
* Will not start any new tinnitus treatment during the study
* Ability to give informed consent and understand study objectives in English
* Willing and able to understand and comply with all study-related procedures

Exclusion Criteria:

* Substantial hearing loss or hyperacusis that may interfere with the study
* Medical history of other ear or brain disorders, history of seizures, or currently using any medication or treatments that can cause or increase the chances of seizures
* Any implanted medical or metal device, such as a pacemaker, aneurysm clip, or cochlear implant
* Pregnant or currently breast-feeding (we need to give all female subjects a pregnancy test because pregnant females and unborn children need extra protection for their safety)
* Any handicap that prevents the subject from reliably performing the tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Change in Tinnitus Functional Index Questionnaire Score | Change from baseline score at 1 week after testing paradigm
  A series of questions to assess the quality and bothering nature of the tinnitus, which is then quantified into a single score.
Change in Minimal Masking Level | Change in baseline level at an expected average of 1 minute and 1.5 hours after testing paradigm
  A narrowband noise (from 2-12 kHz) is presented to the tinnitus ear and the minimum sound level (in decibel sound pressure level, decibel SPL) is determined that completely masks the tinnitus percept.

SECONDARY OUTCOMES:
Change in Tinnitus Handicap Inventory Questionnaire Score | Change from baseline score at 1 week after testing paradigm
  A series of questions to assess the quality and bothering nature of the tinnitus, which is then quantified into a single score.
Change in Tinnitus Rating (0-10, 10 being worst) | Change in baseline rating at an expected average of 4 minutes and 1.5 hours after testing paradigm
  The subject rates the disturbance or bothering nature of the tinnitus.
Change in Tinnitus Subjective Description | Change in baseline description at an expected average of 5 minutes and 1.5 hours after testing paradigm
  The subject describes the quality, characteristics and bothering nature of the tinnitus.
Change in Tinnitus Matching (pitch and loudness) | Change in baseline pitch and loudness at an expected average of 1.5 hours after testing paradigm
  The subject adjusts the loudness and pitch (i.e., frequency) of a sound played to an ear to that of the tinnitus percept.
Daily Tinnitus Journal Entries | 0, 1, 2, 3, 4, 5, 6, 7 days post-testing paradigm
  The subject describes the quality, characteristics and bothering nature of the tinnitus on a daily basis. The subject can also include any unusual or interesting events relating to the tinnitus that he/she feels would be relevant for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Lim, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Nils Hasselmo Hall, 6-105, Minneapolis, Minnesota, United States